CLINICAL TRIAL: NCT04393077
Title: Emotional Freedom Technique (EFT) Effect on Nurses' Stress, Anxiety and Burnout Levels During the COVID-19 Pandemic Process: A Randomized Controlled Study
Brief Title: Emotional Freedom Technique (EFT) Effect on Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Assistant Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020\0192
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Stress; Anxiety; Burnout, Caregiver
Keywords: COVID-19; Emotional Freedom Technique
MeSH Terms: conditions — Anxiety Disorders; Caregiver Burden; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will complete the pre-tests of the introductory features form, SUD, STAI-I, and burnout scales sent via Survey Monkey. The participants (n=40) will be given 15 minutes of free time and asked to be in a position where the individuals were comfortable, in the quietest and most tranquil environment possible. At the end of this period, post-test SUD, STAI-I, and burnout scales will be sent to the participants and they will be asked to fill in the scores.
- Intervention (Experimental): Firstly, people in the entire group fill out the introductory features form on the online questionnaire form. The time of the meeting will be determined by collaborating with the participants in the experimental group. During the interview, they will be asked to be in a position that was comfortable for the individuals, in the quietest and calm environment possible. At the beginning of the meeting, they will be asked to fill in the pre-test SUD, STAI-I, and burnout scales sent via SurveyMonkey. Then, the EFT session (20 minutes) will be conducted once mutually with the researcher, who is an expert in their field. At the end of the session, they will be filled the post-test SUD, STAI-I and burnout scales
  Interventions: Behavioral: Emotional Freedom Technique

INTERVENTIONS:
Behavioral: Emotional Freedom Technique — EFT application was started by showing the meridian points to the participants through the picture. It was advised that these points should be clicked with the index finger and middle finger without hurting, but with certain strokes, and it was ensured that they understood the regions by showing and applying them. Then, the following basic steps, which should be followed by the EFT session (four in total lasting 20 minutes), were carried out in succession with the researcher.
  Arms: Intervention

SUMMARY:
Background: Infectious disease outbreaks have a psychological effect on the general population, and especially on health workers. Nurses who care for COVID-19 patients feel negative emotions, fear, and anxiety due to fatigue, discomfort, and helplessness due to high-intensity work.

Objective: The study aims to evaluate the effect of EFT in the prevention of stress, anxiety, and burnout of nurses who have an important position in the fight against COVID-19.

Design: Randomized controlled trial. Setting: COVID-19 department of a university hospital in Istanbul Province, Turkey.

Participants: The sample of the study consisted of nurses working on 80 COVID-19 cases.

Methods: The investigators will recruit nurses who care for the patient infected with COVID-19 randomly allocated them to the intervention (n = 40) and control (n = 40) groups. EFT will apply to the experimental group with online access. Data will collect using the Introductory Characteristics Form, the Subjective Discomfort Unit Scale, the State-Trait Anxiety Inventory, and the Burnout Scale.

DETAILED DESCRIPTION:
With the onset of the COVID-19 epidemic, healthcare workers have assumed important responsibilities in the control, prevention, care, and treatment of its spread. In this period, they provided the necessary health practices for suspicious or confirmed COVID-19 patients in the front lines and under harsh conditions, which are generally long and tiring. It is clear that infectious disease outbreaks have a psychological effect on the general population, and especially on health workers. The social distance required to prevent outbreaks is a key factor in disease management while causing social and psychological effects.

2.1. Design A randomized controlled experimental research design. The study complied with the guidelines of the Consolidated Standards of Reporting Trials (CONSORT) checklist.

2.2. Participants This study will conduct with nurses working in a university hospital located in Istanbul between May 2020 and June 2020, working in the care of COVID-19 patients.

2.5. Measures The data will be collected with the Introductory Characteristics Form, the positive units of distress scale, the State-Trait Anxiety Inventory, and the Burnout Inventory. The investigators created our data collection forms using Survey Monkey, which provides electronic self-access and prevents data from multiple entries from the same person, making it easier to collect and track data. Confidentiality will be guaranteed by completely disabling electronic and IP address records to obtain anonymous replies.

ELIGIBILITY:
Inclusion Criteria:

* Not taking any courses about coping with anxiety and stress,
* Volunteering to participate in the study.

Exclusion Criteria:

* Having any psychiatric diagnoses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
The subjective units of distress scale | Immediately after EFT implementation
  The cognitive element of EFT involves self-rating of distress severity and pairing of an abbreviated exposure statement and a self-acceptance statement. The severity of distress was evaluated by subjects on an 11-point Likert scale. 0 corresponds to absolutely no distress, while 10 corresponds to the maximum possible distress. This was considered as the subjective units of distress scale (SUD) and provides clinicians and patients with the measurement of the severity of symptoms experienced by the latter in addition to a repeated measure by which the progress can be evaluated.
The State Anxiety | Immediately after EFT implementation
  The State-Trait Anxiety Inventory includes two separate scales with a total of 40 items. This study employed the State Anxiety Scale. Its validity and reliability in Turkish were confirmed by Öner and Lecompte. The scale consists of 20 questions and anxiety questions. To obtain the anxiety scale, to state how the person feels at any time and under any circumstances, answers were requested taking into account the feelings related to the situation.
Burnout | Immediately after EFT implementation
  The scale was created to measure the professional burnout levels of individuals. Adaptation studies in Turkish were carried out by Çapri in (2006) This 7-point Likert type scale consists of 21 items, scoring between 1 (never) and 7 (always), while 4 items (3, 6, 19, 20) of the scale are scored in reverse. While evaluating the scale scores, the increase in the score obtained indicates that burnout increases and the decrease in score indicates that burnout decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Dinçer, Study Chair — Istanbul Medeniyet University
Locations (1):
- Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun N, Wei L, Shi S, Jiao D, Song R, Ma L, Wang H, Wang C, Wang Z, You Y, Liu S, Wang H. A qualitative study on the psychological experience of caregivers of COVID-19 patients. Am J Infect Control. 2020 Jun;48(6):592-598. doi: 10.1016/j.ajic.2020.03.018. Epub 2020 Apr 8. PMID 32334904
- [Background] Hersch RK, Cook RF, Deitz DK, Kaplan S, Hughes D, Friesen MA, Vezina M. Reducing nurses' stress: A randomized controlled trial of a web-based stress management program for nurses. Appl Nurs Res. 2016 Nov;32:18-25. doi: 10.1016/j.apnr.2016.04.003. Epub 2016 Apr 9. PMID 27969025